CLINICAL TRIAL: NCT04160286
Title: The Danish Neuropsychological Study of the Adverse Effects of ECT
Acronym: DANSECT
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Poul Videbech, Professor, consultant in psychiatry, University of Copenhagen
Other Study IDs: DANSECT
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2023-02

CONDITIONS: Depressive Disorder; Depression; Cognitive Dysfunction; Electroconvulsive Therapy
Keywords: Hippocampus; Depression; Electroconvulsive therapy; Brain-Derived Neurotrophic Factor; Magnetic Resonance Imaging; Autobiographical memory; Cognitive side-effects
MeSH Terms: conditions — Depressive Disorder; Depression; Cognitive Dysfunction | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, urine samples and hair samples are kept in the biobank until the last enrolled patient has been examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ECT: Group of patients receiving ECT during their hospitalization.
  Interventions: Other: Electroconvulsive therapy
- Non-ECT: Group of patients not receiving ECT during their hospitalization.
- Healthy controls: Group of healthy participants.

INTERVENTIONS:
Other: Electroconvulsive therapy — Electroconvulsive therapy is a procedure, done under general anesthesia, in which small electric currents are passed through the brain, intentionally triggering a brief seizure.
  Repeated as deemed needed by the patients' doctor. Typically prescribed 10 times (3 times pr week)
  Groups: ECT

SUMMARY:
The main purpose of this study is to investigate the adverse cognitive side-effects of electroconvulsive therapy (ECT). The second aim is to investigate the mechanisms of effect of ECT.

DETAILED DESCRIPTION:
ECT has been the most effective treatment of depression for decades. Despite of this, neither the mechanism of action or side-effects are fully elucidated. The reason why some patients relapse shortly after remission is still not completely understood. Thus, there is a need to find predictors of the favourable clinical effect, relapse and side-effects. ECT is considered by professionals to be a safe procedure. Additionally, many patients do not consent to this treatment because they fear a permanent loss of memory or that they will contract a brain damage after the completed ECT series. Therefore, it is very important to examine whether ECT might have negative effects on the structure or function of the brain, using state of the art Magnetic Resonance Imaging (MRI) techniques.

DANSECT is a prospective, observational follow-up study with the aim of examining why cognitive side-effects of ECT occur and potentially find predictors for whom they may affect by investigating the ECT-associated cognitive disturbances, structural brain changes and clinical outcomes. Second, DANSECT examines the mechanisms of effect of ECT.

DANSECT comprises an ECT-group (30 patients) and a clinical control group (30 patients). The former consists of patients with depression receiving ECT, and the latter consists of matched patients with depression treated pharmacologically. The examinations will take place at three time-points; before, immediately after ECT or just before discharge, and 6 months after. DANSECT is a naturalistic clinical project. This means that the number of ECT sessions given to the patients in the ECT-group is up to the referring physician.

The aim of DANSECT is to investigate the cognitive side-effects of ECT. Specifically, the research project aims to examine:

1. Prevalence, extent and persistence of adverse cognitive effects following ECT.
2. Associations between neuroimaging findings and cognitive changes following ECT.
3. Predictors of adverse cognitive effects of ECT.

Hypotheses:

1. Consistency in autobiographical memories will be reduced over time in both study groups. However, the reduction will be significantly larger for the ECT patients after ECT compared to the control group. The group difference is expected to be present at both short-term and long-term.
2. Autobiographical memory deterioration is expected to correlate with volumetric changes of the hippocampi.
3. Processing speed, anterograde memory and executive functions will be temporarily deteriorated after ECT. The cognitive changes will correlate with volumetric brain changes and changes in structural connectivity.
4. Baseline atrophy, age, years of education and cognitive reserve will predict the cognitive side-effects following ECT.
5. Machine learning will reveal patterns and inference enabling the development of a predictive model of clinical and cognitive outcome after treatment with ECT, by combining neuropsychological tests, structural and functional neuroimaging (MRI) and other neurobiological measures.

In addition, the aim of DANSECT is to investigate the mechanisms of effect of ECT. The secondary aims of the project are thus to examine:

1. Clinical, biochemical and neurobiological predictors of response to ECT
2. Clinical, biochemical and neurobiological predictors of relapse of depression after ECT
3. Biochemical and neurobiological mechanisms of response to ECT

Hypotheses:

1. Smaller baseline hippocampal volume is associated with a larger post-pre reduction of depressive symptoms
2. Thinner cortical thickness predicts better clinical improvement
3. The cortisol trajectory before ECT is associated with clinical outcome
4. Elevated peripheral baseline VEGF is associated with a larger post-pre reduction of depressive symptoms
5. Baseline microRNA levels are associated with clinical outcome
6. A higher baseline structural connectivity predicts better clinical improvement
7. A larger post-ECT increase in hippocampal volume, cortical thickness, BDNF and VEGF predicts a lower risk of relapse within six months after an ECT series

ELIGIBILITY:
Inclusion Criteria:

* age 18-95 years
* admitted at the MHC Glostrup, MHC Amager or MHC Copenhagen (or other Mental Health Centres in the Capital Region)
* fulfilling the criteria for depression according to ICD-10 and where ECT is planned.
* must be able to give informed consent to participate in the study

Exclusion Criteria:

* Schizophrenia or any other psychotic disorder except for psychotic depression
* Dependency syndrome according to ICD-10.
* Severe somatic or neurological condition (e.g. stroke) confounding results
* Head trauma resulting in unconsciousness for more than 5 minutes
* Severe psychotic symptoms or suicide impulses making transportation hazardous
* Contraindications against MRI
* Pregnancy
* Maintenance ECT or ECT received during the last 6 months
* Any form of compulsory treatment
* Subjects who do not consent to be informed of incidental findings that could have healthcare implications will not be scanned and can thus not be included

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of two groups of inpatients admitted to one of the recruiting Mental Health Centres (MHC) in the Capital Region of Denmark, diagnosed with depression according to the 10th version of the International Classification of Diseases (ICD-10) and scheduled to ECT series. Patients in the other group does not received ECT and is thus a control group.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Columbia Autobiographical Memory Interview - Short Form | at baseline (before ECT series)
  Measures consistency in autobiographical memories over time. Scoring: Minimum: 0. Maximum: 60. A higher score means a better cognitive performance.
Columbia Autobiographical Memory Interview - Short Form | at 5 (+/- 2) days after completion of the ECT series
  Measures consistency in autobiographical memories over time. Scoring: Minimum: 0. Maximum: 60. A higher score means a better cognitive performance.
Columbia Autobiographical Memory Interview - Short Form | at follow-up (6 (+/-2) months after the ECT series
  Measures consistency in autobiographical memories over time. Scoring: Minimum: 0. Maximum: 60. A higher score means a better cognitive performance.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Hamilton Depression Rating Scale 6-item. Scoring: Minimum: 0. Maximum: 22. A higher score means more symptom severity.
The Screen for Cognitive Impairment for Psychiatry | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Screening tool to measure cognitive performance across several cognitive domains. Scoring: Minimum 0. Maximum: Unlimited. A higher score means a better cognitive performance.
Reys complex figure task | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures visuospatial, constructional, executive and anterograde memory abilities. Scoring: Minimum: 0. Maximum: 36. A higher score means a better cognitive performance.
Trail Making Test A | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures psychomotor speed. Scoring: Minimum:0. Maximum: Unlimited. A higher score means a worse cognitive performance.
Trail Making Test B | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures complex psychomotor speed / executive function. Scoring: Minimum:0. Maximum: Unlimited. A higher score means a worse cognitive performance.
Digit span (WAIS-IV) | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures attention span (forwards) and working memory (backwards). Scoring: Minimum: 0. Maximum: 16.
Five Point Test | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures spatial fluency / problem solving. Scoring: Minimum: 0. Maximum: Unlimited. A higher score means a better cognitive performance.
Color-Word Interference Test (D-KEFS) | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures psychomotor speed, meantal flexibility and set-shifting. Scoring: Minimum: 0. Maximum: Unlimited. A higher score means a worse cognitive performance.
Symbol Digit Modalities Test | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures psychomotor speed. Scoring: Minimum: 0. Maximum: Unlimited. A higher score means a worse cognitive performance.
Vividness of Visual Imagery Questionnaire - Danish version | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Measures subjective experience of the vividness of ones mental visual imagery. Scoring: Minimum: 16. Maximum: 80. A higher score means more vividly experienced mental imagery.
Vocabulary (WAIS-IV) | at one time point: at 5 (+/- 2) days after completion of the ECT series
  Measures vocabulary and serves as an estimate of premorbid intellectual ability. Scoring: Minimum: 0. Maximum: 57. A higher score means a better vocabulary.
Cognitive complaints in bipolar disorder rating assessment | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Self-report of experienced cognitive difficulties. Scoring: Minimum: 0. Maximum: 48. A higher score means more symptom severity.
Squire Subjective Memory Questionnaire | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Self-report of experienced memory difficulties. Scoring: Minimum: -72. Maximum: +72. A higher score means a better cognitive function.
Paired Associates Learning (CANTAB) | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Visuospatial pattern localization. Scoring: Minimum 0. Maximum: Unlimited. A higher score (errors) means a worse cognitive performance.
WHO-5 | at 3 time points: at baseline (before ECT series), at 5 (+/- 2) days after completion of the ECT series, at follow-up (6 (+/-2) months after the ECT series)
  Self-report of well-being in the last 14 days. Scoring: Minimum: 0. Maximum: 25. A higher score means a better experience of well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Poul Videbech, Professor, Principal Investigator — University of Copenhagen & Mental Health Centre Glostrup
Locations (1):
- Mental Health Services of the Capital Region of Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Patient Data.

REFERENCES:
- [Background] Abbott CC, Gallegos P, Rediske N, Lemke NT, Quinn DK. A review of longitudinal electroconvulsive therapy: neuroimaging investigations. J Geriatr Psychiatry Neurol. 2014 Mar;27(1):33-46. doi: 10.1177/0891988713516542. Epub 2013 Dec 30. PMID 24381234
- [Background] Andrade C, Bolwig TG. Electroconvulsive therapy, hypertensive surge, blood-brain barrier breach, and amnesia: exploring the evidence for a connection. J ECT. 2014 Jun;30(2):160-4. doi: 10.1097/YCT.0000000000000133. PMID 24800688
- [Background] Ahdidan J, Hviid LB, Chakravarty MM, Ravnkilde B, Rosenberg R, Rodell A, Stodkilde-Jorgensen H, Videbech P. Longitudinal MR study of brain structure and hippocampus volume in major depressive disorder. Acta Psychiatr Scand. 2011 Mar;123(3):211-9. doi: 10.1111/j.1600-0447.2010.01644.x. Epub 2011 Jan 11. PMID 21219263
- [Background] Arts B, Peters M, Ponds R, Honig A, Menheere P, van Os J. S100 and impact of ECT on depression and cognition. J ECT. 2006 Sep;22(3):206-12. doi: 10.1097/01.yct.0000235925.37494.2c. PMID 16957538
- [Background] Awata S, Konno M, Kawashima R, Suzuki K, Sato T, Matsuoka H, Fukuda H, Sato M. Changes in regional cerebral blood flow abnormalities in late-life depression following response to electroconvulsive therapy. Psychiatry Clin Neurosci. 2002 Feb;56(1):31-40. doi: 10.1046/j.1440-1819.2002.00927.x. PMID 11929569
- [Background] Bergsholm P, Larsen JL, Rosendahl K, Holsten F. Electroconvulsive therapy and cerebral computed tomography. A prospective study. Acta Psychiatr Scand. 1989 Dec;80(6):566-72. doi: 10.1111/j.1600-0447.1989.tb03027.x. PMID 2618780
- [Background] Beyer JL. Volumetric brain imaging studies in the elderly with mood disorders. Curr Psychiatry Rep. 2006 Feb;8(1):18-24. doi: 10.1007/s11920-006-0077-0. PMID 16513039
- [Background] Bolwig TG, Hertz MM, Paulson OB, Spotoft H, Rafaelsen OJ. The permeability of the blood-brain barrier during electrically induced seizures in man. Eur J Clin Invest. 1977 Apr;7(2):87-93. doi: 10.1111/j.1365-2362.1977.tb01578.x. PMID 404164
- [Background] Bolwig TG. How does electroconvulsive therapy work? Theories on its mechanism. Can J Psychiatry. 2011 Jan;56(1):13-8. doi: 10.1177/070674371105600104. PMID 21324238
- [Background] Bolwig TG. Neuroimaging and electroconvulsive therapy: a review. J ECT. 2014 Jun;30(2):138-42. doi: 10.1097/YCT.0000000000000140. PMID 24800687
- [Background] Bronge L, Wahlund LO. White matter changes in dementia: does radiology matter? Br J Radiol. 2007 Dec;80 Spec No 2:S115-20. doi: 10.1259/bjr/35265137. PMID 18445741
- [Background] Brunoni AR, Baeken C, Machado-Vieira R, Gattaz WF, Vanderhasselt MA. BDNF blood levels after electroconvulsive therapy in patients with mood disorders: a systematic review and meta-analysis. World J Biol Psychiatry. 2014 Jul;15(5):411-8. doi: 10.3109/15622975.2014.892633. Epub 2014 Mar 16. PMID 24628093
- [Background] Campbell JJ 3rd, Coffey CE. Neuropsychiatric significance of subcortical hyperintensity. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):261-88. doi: 10.1176/jnp.13.2.261. No abstract available. PMID 11449035
- [Background] Coffey CE, Weiner RD, Djang WT, Figiel GS, Soady SA, Patterson LJ, Holt PD, Spritzer CE, Wilkinson WE. Brain anatomic effects of electroconvulsive therapy. A prospective magnetic resonance imaging study. Arch Gen Psychiatry. 1991 Nov;48(11):1013-21. doi: 10.1001/archpsyc.1991.01810350053008. PMID 1747016
- [Background] Dukart J, Regen F, Kherif F, Colla M, Bajbouj M, Heuser I, Frackowiak RS, Draganski B. Electroconvulsive therapy-induced brain plasticity determines therapeutic outcome in mood disorders. Proc Natl Acad Sci U S A. 2014 Jan 21;111(3):1156-61. doi: 10.1073/pnas.1321399111. Epub 2013 Dec 30. PMID 24379394
- [Background] Fitzgerald PB, Laird AR, Maller J, Daskalakis ZJ. A meta-analytic study of changes in brain activation in depression. Hum Brain Mapp. 2008 Jun;29(6):683-95. doi: 10.1002/hbm.20426. PMID 17598168
- [Background] UK ECT Review Group. Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003 Mar 8;361(9360):799-808. doi: 10.1016/S0140-6736(03)12705-5. PMID 12642045
- [Background] Herrmann LL, Le Masurier M, Ebmeier KP. White matter hyperintensities in late life depression: a systematic review. J Neurol Neurosurg Psychiatry. 2008 Jun;79(6):619-24. doi: 10.1136/jnnp.2007.124651. Epub 2007 Aug 23. PMID 17717021
- [Derived] Mathiassen AB, Lundsgaard CC, Gbyl K, Miskowiak K, Fagerlund B, Larsson HBW, Lindberg U, Videbech P. Brain reserve in memory regions is associated with the preservation of autobiographical memories after electroconvulsive therapy. Front Psychiatry. 2025 Nov 10;16:1699102. doi: 10.3389/fpsyt.2025.1699102. eCollection 2025. PMID 41293195
- See also: Danish Health Authority: Reference Programme for Treating Unipolar Depression in adults. 2007. — http://www.sst.dk/~/media/6F9CE14B6FF245AABCD222575787FEB7.ashx